CLINICAL TRIAL: NCT01967498
Title: Montelukast for Children With Chronic Otitis Media With Effusion (COME): A Double-blind, Placebo-controlled Study
Acronym: COME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-13-MH-0170-13-CTIL
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Otitis Media With Effusion; Conductive Hearing Loss
Keywords: chronic otitis media with effusion; conductive hearing loss
MeSH Terms: conditions — Hearing Loss, Conductive | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- montelukast (Experimental): this arm will receive montelukast as the active intervention of the study
  Interventions: Drug: Montelukast
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Montelukast
  Other Names: Singulair
  Arms: montelukast

SUMMARY:
The purpose of our double-blind, placebo controlled study is to test the hypothesis that montelukast therapy might be associated with improved hearing in certain sub populations of children suffering from OME.

DETAILED DESCRIPTION:
Chronic otitis media with effusion is a common problem in children that sometimes causes hearing impairment which may affect language development and quality of life of the child. The standard treatment is surgical insertion of ventilation tubes. In the pediatric population this procedure is preformed under general anesthesia and is associated with quite a few possible complications.

In this study we will examine the effects of conservative treatment with montelukast on the resolution of the effusion without surgical treatment .

Montelukast is a selective leukotriene receptor antagonist that is widely used for children with asthma1. Allergic rhinitis in children is one of the approved indications for Montelukast.

Montelukast's effect on OME has been studied in several previous studies. In 2004 a study by Combs JT2 showed efficacy of 49% of Montelukast in clearing persistent OME post-AOM. This study was not directed at patients with chronic OME and did not use audiometry as an endpoint. Another study from 2005 by Balatsouras DG studied the effect of montelukast on OME in children suffering from co-existing asthma. The rate of OME resolution after one month of treatment was 60% as opposed to 36% in the control group. The endpoint of this study was OME and not audiometry results. There was no additional followup. In 2010 Schoem SR began a randomized control double blinded study testing the effect of montelukast on children with confirmed OME of 2 months. Montelukast was given for one month. Although the goal was to recruit 120 children, the study was halted after 38 were treated because a statistical trend showed that there was no positive effect compared to the placebo group.

An additional study was published in 2007 performed as a RCT of 77 children did not prove the drug's effectiveness as a treatment for OME . This study was published as an abstract only and no details of the hearing or inclusion criteria were given. Montelukast has been proven effective in resolving experimental OME in a rat model although as opposed to methylpresnisone it did not reduce the submucosal neutrophil infiltrate.

The purpose of our double-blind, placebo controlled study is to test the hypothesis that montelukast therapy might be associated with improved hearing in certain sub populations of children suffering from OME.

ELIGIBILITY:
Inclusion Criteria:

* Documented persistent OME of at least 3 months (otoscopy or audiometry or tympanometry)
* Patients between the ages of 2-10 being evaluated for VT surgery
* Tympanogram type B
* A conductive hearing loss greater than 20 DB
* Otoscopy confirming middle ear effusion

Exclusion Criteria:

* previous adenoidectomy or tonsillectomy
* history of ear surgery
* cleft palate, Down's syndrome, congenital, malformations of the ear or cholesteatoma
* Sensoneural hearing loss
* Allergy to montelukast
* Moderate or Severe OSA requiring surgery sooner than 3 months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
improvement of hearing of 10 db based on pure tone audiometry | 3 months

SECONDARY OUTCOMES:
improvement of tympanometry graph to type A | 3 months